CLINICAL TRIAL: NCT01340625
Title: A Relative Bioavailability Study of 0.4 mg/35 Mcg Norethindrone and Ethinyl Estradiol Chewable Tablets Under Fasting Conditions
Brief Title: Norethindrone/Ethinyl Estradiol 0.4 mg/35 Mcg Chewable Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: R06-1188
Record Dates: First submitted 2011-04-20; First posted 2011-04-22 (Estimated); Results first posted 2011-05-25 (Estimated); Last update posted 2011-05-25 (Estimated); Status verified 2011-04

CONDITIONS: Bioequivalence
Keywords: Healthy Subjects
MeSH Terms: interventions — ovcon 35; Norethindrone; Ethinyl Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Investigational Test Product (Experimental): Norethindrone/Ethinyl Estradiol 0.4 mg/35 mcg Chewable Tablets (Teva)
  Interventions: Drug: Norethindrone/Ethinyl Estradiol
- Reference Listed Drug (Active Comparator): Ovcon® 35 Fe 0.4 mg/35 mcg Chewable Tablets (Warner Chilcott)
  Interventions: Drug: Ovcon® 35 Fe

INTERVENTIONS:
Drug: Norethindrone/Ethinyl Estradiol — 0.4 mg/35 mcg Chewable Tablets
  Other Names: Zeosa®
  Arms: Investigational Test Product
Drug: Ovcon® 35 Fe — 0.4 mg/35 mcg Chewable Tablets
  Other Names: Femcon® Fe; Norethindrone/Ethinyl Estradiol (generic name)
  Arms: Reference Listed Drug

SUMMARY:
This study compared the relative bioavailability (rate and extent of absorption) of 0.4 mg/35 mcg Norethindrone and Ethinyl Estradiol Chewable Tablets by Teva Pharmaceuticals, USA with that of 0.4 mg/35 mcg Ovcon® 35 Fe Chewable Tablets manufactured by Warner Chilcott Company, Inc., following a single oral dose (2 * 0.4 mg/35 mcg chewable tablets) in healthy female adult volunteers administered under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers who have been informed of the nature of the study and agree to read, review, and sign the informed consent document prior to Period I dosing.
* Volunteers who have completed the screening process within 28 days prior to Period I dosing.
* Volunteers who are healthy adult women 18-35 years of age, inclusive, at the time of dosing.
* Volunteers who have a body mass index (BMI) between 19-30 kg/m2, inclusive, and weight at least 110 lbs.
* Volunteers who are healthy as documented by the medical history, physical examination, vital sign assessments, 12-lead electrocardiogram, clinical laboratory assessments, and by general observations. The physical examination will also include a gynecological exam. If the subject has completed an acceptable Papanicolaou smear and gynecological exam in the previous 12 months and documentation of acceptable results are provided, both will be deferred. Any abnormalities/deviations from the normal range that might be considered clinically relevant by the study physician and investigator will be evaluated for individual cases, documented in study files, and agreed upon by both the study physician and investigator prior to enrolling the volunteer in this study and for continued enrollment.
* Volunteers must practice an acceptable non-hormonal birth control method as judged by the investigator(s) at least 14 days prior to Period I dosing, throughout the study, and until 14 days after second period dosing.

Exclusion Criteria:

* Volunteers who report receiving any investigational drug within 30 days prior to Period I dosing.
* Volunteers who report taking any oral contraceptives including estrogen and progestin combined pills and progestin only pills or patch within 28 days prior to Period I dosing, using injectable contraceptives within 6 months of first period dosing.
* Volunteers who have ever had progestational hormone implants.
* Volunteers who report any presence or history of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic systems or psychiatric disease as determined by the clinical investigator(s).
* Volunteers who report any presence or history of migraines or severe headaches.
* Volunteers who have systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 45 or over 90 mmHg will be excluded from the study.
* Volunteers who have a history of thrombotic disorders or have ever had cerebrovascular accident or transient ischemic attacks.
* Volunteers with a history of breast cancer or undiagnosed breast nodules, active malignancies or undiagnosed vaginal bleeding.
* Volunteers having other conditions that may be aggravated by fluid retention (as determined by principal investigator).
* Volunteers who have a history of jaundice with previous use of oral contraceptives or any other kinds of hormonal contraceptives.
* Volunteers whose clinical laboratory test values fall outside the accepted reference range and when confirmed on re-examination is deemed to be clinically significant.
* Volunteers who demonstrate a reactive screen for hepatitis B surface antigen, hepatitis C antibody, or HIV antibody.
* Volunteers who report a history of allergic response(s) to norethindrone/ethinyl estradiol or progestin/estrogens or related drugs.
* Volunteers who report the use of any systemic prescription medication in the 14 days prior to Period I dosing (with the exception of hormonal contraceptives).
* Volunteers with a history of clinically significant allergies including drug allergies.
* Volunteers who report a clinically significant illness during the 4 weeks prior to Period I dosing (as determined by the clinical investigators).
* Volunteers who report a history of drug or alcohol addiction or abuse within the past year.
* Volunteers who demonstrate a positive drug abuse screen for this study prior to Period I dose administration.
* Volunteers who currently use or have used tobacco products within 30 days prior to Period I dosing.
* Volunteers who report donating greater that 150 mL of blood within 30 days prior to Period I dosing. All subjects will be advised not to donate blood for 4 weeks after completing the study.
* Volunteers who report donating plasma within 30 days prior to Period I dosing. All subjects will be advised not to donate plasma for 4 weeks after completing the study.
* Volunteers who demonstrate a positive pregnancy screen.
* Volunteers who are currently pregnant of breastfeeding.
* Volunteers who are using or have used within the 3 months preceding Period I dosing any vaginally administered estrogen or progestin-containing products.
* Any volunteer who engages in unprotected sexual intercourse during the time interval starting 14 days prior to first period dosing and until 14 days after the Period II dosing.
* Volunteers who have had a hysterectomy or oophorectomy (unilateral or bilateral).

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2006-12; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- PRACS Institute, Ltd., Fargo, North Dakota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Norethindrone/Ethinyl Estradiol (Test) First: 0.4 mg/35 mcg Norethindrone/Ethinyl Estradiol Chewable Tablets test product dosed in first period followed by 0.4 mg/35 mcg Ovcon® 35 Fe Chewable Tablets reference product dosed in the second period.
- Ovcon® 35 Fe (Reference) First: 0.4 mg/35 mcg Ovcon® 35 Fe Chewable Tablets reference product dosed in first period followed by 0.4 mg/35 mcg Norethindrone/Ethinyl Estradiol Chewable Tablets test product dosed in the second period.
Period: First Intervention
Arm/Group | Norethindrone/Ethinyl Estradiol (Test) First | Ovcon® 35 Fe (Reference) First
Started | 18 | 18
Completed | 17 | 18
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Washout Period of 28 Days
Arm/Group | Norethindrone/Ethinyl Estradiol (Test) First | Ovcon® 35 Fe (Reference) First
Started | 17 | 18
Completed | 16 | 18
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Second Intervention
Arm/Group | Norethindrone/Ethinyl Estradiol (Test) First | Ovcon® 35 Fe (Reference) First
Started | 16 | 18
Completed | 16 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Norethindrone/Ethinyl Estradiol (Test) First | Ovcon® 35 Fe (Reference) First | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 18 | 36
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian | 0 | 1 | 1
  Caucasian | 18 | 17 | 35
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Norethindrone
Description: Bioequivalence based on Norethindrone Cmax (maximum observed concentration of drug substance in plasma).
Time Frame: Blood samples collected over a 60 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Norethindrone/Ethinyl Estradiol (Test): 0.4 mg/35 mcg Norethindrone/Ethinyl Estradiol Chewable Tablets test product dosed in either period.
- Ovcon® 35 Fe (Reference): 0.4 mg/35 mcg Ovcon® 35 Fe Chewable Tablets reference product dosed in either period.
Arm/Group | Norethindrone/Ethinyl Estradiol (Test) | Ovcon® 35 Fe (Reference)
Number analyzed (Participants) | 34 | 34
ng/mL | 10.94 (5.22) | 10.00 (4.13)
Statistical Analysis 1: Comparison: Norethindrone/Ethinyl Estradiol (Test) vs Ovcon® 35 Fe (Reference); Test type: Non-Inferiority or Equivalence — ANOVA is to be used to identify the source contributions by factors including subjects, period, formulation and potential interactions. The geometric mean ratio together with the ANOVA residual mean error term are used to identify the statistical basis for the 90% confidence interval for the ratio of the population means (Test [T]/Reference[R]) of the identified metrics (e.g. AUC, Cmax); Ratio of the T/R geometric mean x 100 = 107.84, 90% CI 2-sided [100.91 to 115.24] — Bioequivalence is established if the 90% confidence interval for the ln-transformed geometric mean between the reference (R) and test (T) product fall within the interval of 80-125%

2. Primary Outcome: AUC0-t of Norethindrone
Description: Bioequivalence based on Norethindrone AUC0-t (area under the concentration-time curve from time zero to time of last measurable concentration).
Time Frame: Blood samples collected over a 60 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Norethindrone/Ethinyl Estradiol (Test) | Ovcon® 35 Fe (Reference)
Number analyzed (Participants) | 34 | 34
ng*h/mL | 43.83 (30.50) | 40.73 (22.41)
Statistical Analysis 1: Comparison: Norethindrone/Ethinyl Estradiol (Test) vs Ovcon® 35 Fe (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 104.03, 90% CI 2-sided [96.74 to 111.88] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: AUC0-inf of Norethindrone
Description: Bioequivalence based on Norethindrone AUC0-inf (area under the concentration-time curve from time zero to infinity).
Time Frame: Blood samples collected over a 60 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Norethindrone/Ethinyl Estradiol (Test) | Ovcon® 35 Fe (Reference)
Number analyzed (Participants) | 34 | 34
ng*h/mL | 48.67 (34.36) | 45.43 (27.03)
Statistical Analysis 1: Comparison: Norethindrone/Ethinyl Estradiol (Test) vs Ovcon® 35 Fe (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 101.97, 90% CI 2-sided [95.73 to 108.62] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Cmax of Ethinyl Estradiol
Description: Bioequivalence based on Ethinyl Estradiol Cmax (maximum observed concentration of drug substance in plasma).
Time Frame: Blood samples collected over a 60 hour period.
Population: 34 out of 36 subjects completed the study. Subjects 13 & 35 were excluded from the statistical analysis for Ethinyl Estradiol due to pre-dose concentrations greater than 5% of Cmax; therefore analysis included 32 data sets.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Norethindrone/Ethinyl Estradiol (Test) | Ovcon® 35 Fe (Reference)
Number analyzed (Participants) | 32 | 32
pg/mL | 230.56 (74.02) | 237.00 (62.90)
Statistical Analysis 1: Comparison: Norethindrone/Ethinyl Estradiol (Test) vs Ovcon® 35 Fe (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 96.24, 90% CI 2-sided [90.04 to 102.86] — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: AUC0-t of Ethinyl Estradiol
Description: Bioequivalence based on Ethinyl Estradiol AUC0-t (area under the concentration-time curve from time zero to time of last measurable concentration).
Time Frame: Blood samples collected over a 60 hour period.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Norethindrone/Ethinyl Estradiol (Test) | Ovcon® 35 Fe (Reference)
Number analyzed (Participants) | 32 | 32
pg*h/mL | 1976.72 (518.96) | 1989.82 (475.30)
Statistical Analysis 1: Comparison: Norethindrone/Ethinyl Estradiol (Test); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 98.80, 90% CI 2-sided [93.89 to 103.97] — [estimate comment as in outcome 1, analysis 1]

6. Primary Outcome: AUC0-inf of Ethinyl Estradiol
Description: Bioequivalence based on Ethinyl Estradiol AUC0-inf (area under the concentration-time curve from time zero to infinity).
Time Frame: Blood samples collected over a 60 hour period.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Norethindrone/Ethinyl Estradiol (Test) | Ovcon® 35 Fe (Reference)
Number analyzed (Participants) | 32 | 32
pg*h/mL | 2129.43 (560.04) | 2131.84 (545.91)
Statistical Analysis 1: Comparison: Norethindrone/Ethinyl Estradiol (Test) vs Ovcon® 35 Fe (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 99.59, 90% CI 2-sided [94.91 to 104.50] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the course of the study, which was approximately 6 weeks in duration.
Description: Volunteers were monitored throughout the study for any adverse experiences. AEs were collected through both solicited and unsolicited methods. The volunteers were encouraged to report signs, symptoms, and any changes in health to the clinic staff.
Arm/Group | Norethindrone/Ethinyl Estradiol (Test) First | Ovcon® 35 Fe (Reference) First
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 14/36 | 12/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Norethindrone/Ethinyl Estradiol (Test) First (N=36) | Ovcon® 35 Fe (Reference) First (N=36)
Diarrhoea (General disorders) | 0 (0) | 2 (2)
Headache (General disorders) | 9 (11) | 9 (11)
Nausea (General disorders) | 8 (9) | 1 (2)
Pallor (General disorders) | 2 (2) | 0 (0)
Syncope (General disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator is not permitted to discuss or publish trial results.